CLINICAL TRIAL: NCT01832428
Title: A Clinical Trial to Study the Safety and Efficacy of Bone Marrow Derived Autologous Cell for the Treatment of Stroke. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: A Clinical Trial to Study the Safety and Efficacy of Bone Marrow Derived Autologous Cell for the Treatment of Stroke.
Acronym: BMACS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00107
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Stroke,
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transfer of autologous MNC intrathecally (Other): Intra thecal transplantation of autologous stem cells 100 Millions per dose in 3 divided doses at interval of 7days.
  Interventions: Other: Intra thecal transplantation of Autologous Stem Cells

INTERVENTIONS:
Other: Intra thecal transplantation of Autologous Stem Cells — Intra thecal transplantation of Autologous Stem Cells

SUMMARY:
This study is single, centre trial to study the safety and efficacy of Bone marrow derived autologous MNCS(100 million per dose)trial to be conducted for 36 months in stroke patients , the primary outcome measure will be the improvement in muscle power of Body and face

DETAILED DESCRIPTION:
This study is single centre trial to study the safety and efficacy of Bone marrow derived autologous MNCS(100 million per dose)trial to be conducted for 36 months in stroke patients , the primary outcome measure will be the improvement in muscle power of Body and face

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from stroke due to cerebral infarct or Haemorrhage or accelerated hypertension.
* willingness to undergo bone marrow derived autologous cell therapy.
* patient those provide fully Informed consent form for the study.
* Ability and willingness to regular visit to hospital and follow up during the protocol Procedure.

Exclusion Criteria:

* Patients with pre - existing or Current systemic disease such as lung , liver ( exception; History of uncomplicated Hepatitis A),gastrointestinal, Cardiac , Immunodeficiency,(including HIV) Or laboratory Investigation that could cause a neurological defect.History of Life threating Allergic or immune- mediated reaction.
* Alcohol and drug abuse / dependence.
* Severe skin infection.
* Haemodynamically unstable.
* subject with primary and secondary diabetes , Insulin depenence,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in power of Body and facial Muscles | 6 Months
  Improvement in power of Body and facial Muscles.

SECONDARY OUTCOMES:
Improvement in Walking Ability | 6 months
  Improvement in Walking Ability in 6 month.
Improvement In Speech and cognition | 6 Months
  - Improvement In Speech and cognition ,Time period-6 month
Improvement in Vision in both eyes | 6 month
  Improvement in Vision in both eyes 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India